CLINICAL TRIAL: NCT05833217
Title: Obesity, Insulin Resistance, and PASC: Persistent SARS-CoV-2 Infection and Inflammation in Human Adipose Tissue
Brief Title: Obesity, Insulin Resistance, and PASC: Persistent SARS-CoV-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Tracey McLaughlin, Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 69063
Record Dates: First submitted 2023-04-26; First posted 2023-04-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Long COVID; Insulin Resistance; Insulin Sensitivity
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Chart Review (not actively recruiting) (No Intervention): Chart review of previously consented participants from the entire NIH RECOVER cohort, comprised of 15,000 infected and 2,600 noninfected patients across the country.
- COVID infected and healthy controls (Experimental): Participants will perform a needle fat biopsy for tissue harvesting in the subacute phase (15-30d) of Covid-19 infection or as a healthy control. Our goal is 20 COVID-19 infected participants and 10 healthy controls.
  Interventions: Procedure: Adipose Tissue Biopsy
- Healthy Controls Only (Experimental): We are looking for 20 healthy controls for 2 in-person visits on separate days.
  1. An Insulin Sensitivity Test (SSPG: Steady State Plasma Glucose) is performed to determine if the participant is insulin-sensitive or insulin resistant.
  2. A Needle Fat Biopsy: After an overnight fast, approximately 1-2 grams of subcutaneous fat will be removed by a needle. Patients will have a local anesthetic prior to the procedure.
  Interventions: Procedure: Adipose Tissue Biopsy; Diagnostic Test: Steady State Plasma Glucose (SSPG) Test

INTERVENTIONS:
Procedure: Adipose Tissue Biopsy — After an overnight fast, approximately 1-2 grams of subcutaneous fat will be removed by a needle. Participants will have a local anesthetic prior to the procedure. The needle fat biopsy will be repeated at quarterly intervals for one year (every 3 months). We will also draw 1 10mL tube of blood at each biopsy for measurement of inflammatory cytokines.
  Arms: COVID infected and healthy controls; Healthy Controls Only
Diagnostic Test: Steady State Plasma Glucose (SSPG) Test — An Insulin Sensitivity Test (SSPG: Steady State Plasma Glucose) is performed to determine if participants are insulin sensitive or insulin resistant. This test is approximately 5-6 hours in length. Participants will be asked to fast for 12 hours. The insulin sensitivity test is designed to measure how well your cells remove glucose from your blood in response to insulin. During this test participants will have two small catheters (tubing) placed in their veins (I.V. lines). The total amount of blood that will be drawn during this test will be 140 mL of blood (approximately 9.5 tablespoons). Insulin is a natural hormone, and octreotide (a synthetic hormone) is a drug that temporarily blocks the secretion of insulin from your pancreas. A member of the research team is present and monitoring the results along with the nursing staff.
  Other Names: Insulin Sensitivity Test
  Arms: Healthy Controls Only

SUMMARY:
The investigators are studying the pathophysiologic links between obesity, insulin resistance (IR), adipose tissue infection, and post-acute sequelae of COVID-19 (PASC). This study looks at whether adipose (fat) tissue contributes to PASC by driving chronic inflammation or by serving as a reservoir for SARS-CoV-2 persistence. The results will not only determine whether obesity and IR are risk factors for PASC, but will also define fundamental biology that sets the stage for the investigation of novel or existing therapies that target the causal pathways identified.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 80
* BMI ≥ 25 kg/m2
* not currently pregnant

Exclusion Criteria:

Arm 2 (Adipose Tissue Biopsy) exclusions include

* pregnancy
* prior liposuction
* recent change in weight (> 2 kg in one month)
* bleeding disorders
* anticoagulant use

Arm 3 (healthy controls only) exclusions include patients with

* major organ disease
* diabetes
* history of liposuction
* bariatric surgery
* eating disorders
* psychiatric disorders
* pregnancy or lactation
* recent change in weight (over the past 12 weeks),
* use of weight loss medication or oral steroids
* hematocrit < 33%
* fasting glucose >= 126 mg/dL
* blood pressure >160/100 mmHg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-05-02 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Triglyceride/HDL-cholesterol ratio | 2 years
  Investigate the relationship between insulin resistance, as described by triglyceride/HDL-cholesterol ratio, and incident PASC (long COVID).
Concentration of Viral RNA in Adipose Tissue | 2 years
  Investigate the expression of viral RNA in adipose tissue in response to COVID-19 infection. Compare adipose tissue transcripts such as known MODY transcription factors measured by PCR between COVID-19 infected participants and healthy controls.
Rate of Inflammatory Response | 2 years
  Investigate inflammatory response to PPARgamma agonist (drug) and other compounds tested in vitro in human fat cells. Compare plasma inflammatory cytokine levels in serum samples as measured by Luminex immunoassay between participants identified as Insulin Sensitive (IS) and Insulin Resistant (IR) using the 2-stage Steady State Plasma Glucose test.
Rate of Inflammatory Gene Expression in Adipose Tissue | 2 years
  Investigate the expression of inflammatory genes in adipose tissue in response to COVID-19 infection. Compare adipose tissue transcripts such as defensin chemokine receptors and platelet activation factors measured by PCR between COVID-19 infected participants and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey McLaughlin, MD, Principal Investigator — Stanford School of Medicine
Locations (2):
- United States (2):
  - Clinical and Translational Research Unit, Palo Alto, California
  - Stanford Health, Palo Alto, California

IPD SHARING:
Plan to Share IPD: No